CLINICAL TRIAL: NCT00730301
Title: A Multi-Center, Prospective, Clinical Trial Designed to Study the Efficacy of One-Way Valve Implantation Based on a New Treatment Algorithm in Patients With Heterogeneous Emphysema
Brief Title: EUROPT Clinical Trial to Study the Efficacy of One-Way Valve Implantation (New Treatment Algorithm) in Patients With Heterogeneous Emphysema
Acronym: EUROPT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LudwLudwig Boltzmann Institute for COPD and Respiratory Epidemiology (Network)
Responsible Party: Arschang Valipour, M.D., Ludwig Boltzmann Institut for COPD
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EUROPT 07-074-0507
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Emphysema; Chronic Obstructive Pulmonary Disease
Keywords: Emphysema; Chronic obstructive pulmonary disease; Lung volume reduction; Lung function
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive | interventions — Pneumonectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Bronchoscopic Lung Volume Reduction (BLVR) — Procedure under general anesthesia.
  Other Names: ZephyrTM Endobronchial Valve (EBV) (Emphasys Medical, Inc., Redwood City, CA)

SUMMARY:
The purpose of this study is to assess the efficacy of a new treatment algorithm for bronchoscopic lung volume reduction (BLVR) in patients with emphysema based on the information of emphysema heterogeneity, destruction score, and fissure analysis.

DETAILED DESCRIPTION:
Emphysema is a progressive pulmonary disease characterized by abnormal and permanent enlargement of air spaces distal to terminal bronchioles accompanied by the destruction of pulmonary parenchyma. Treatment includes inhaled bronchodilator therapy, rehabilitation and/or oxygen treatment. In addition to the above, patients with severe emphysema may benefit from surgical lung volume reduction and/or lung transplantation. The rationale for lung volume reduction surgery is that reducing lung size would restore elastic recoil of the lung and improve chest wall and diaphragm mechanics. It has previously been shown that particularly patients with heterogeneous emphysema seem to benefit most from surgical lung volume reduction.

Bronchoscopic lung volume reduction (BLVR) has recently been introduced as a less invasive potential alternative to surgical lung volume reduction. BLVR attempts to achieve the effects of surgery, by placing bronchial prostheses using a fibreoptic bronchoscope to selectively occlude the airways supplying the most affected hyperinflated regions of the emphysematous lung, while permitting exhaled gas to escape. This attempts to achieve segmental or lobar volume reduction, simulating the effects of surgical LVR. Recent trials of BLVR using endobronchial one-way valves demonstrated significant improvements in lung function parameters, exercise capacity and quality of life in patients with end-stage emphysema. The treatment algorithm for valve implantations to achieve BLVR, however, varied considerably in these reports as well as clinical and functional response rates. Subset analysis of these studies revealed that particularly, but not exclusively, patients with radiological signs of lung volume reduction treated unilaterally showed significant clinical improvements, whereas most patients without signs of lung volume reduction did not experience these benefits. The present study investigates the response to BLVR based on a new treatment algorithm including lung function criteria and computed tomography of the thorax.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed by HRCT Core Lab with eligible heterogeneous disease distribution and at least one complete oblique fissure.
* Age from 40 to 75 years
* BMI < 32 kg/m2
* FEV1 < 40% of predicted value, FEV1/FVC < 70%
* TLC > 120% predicted, RV > 150% predicted.
* Stable with < 20 mg prednisone (or equivalent) qd
* PaCO2 < 50mm Hg
* PaO2 > 45 mm Hg on room air
* 6-min walk of > 50m (without rehabilitation) or > 100m (with rehabilitation)
* Nonsmoking for 4 months prior to initial interview and throughout screening
* The patient agrees to all protocol required follow-up intervals.
* The patient has no child bearing potential
* The patient is willing and able to complete protocol required baseline assessments and procedures

Exclusion Criteria:

* Prior endobronchial treatment for emphysema
* Pleural or interstitial disease that precludes surgery.
* Prior lung transplant, LVRS, median sternotomy, bullectomy or lobectomy.
* Clinically significant bronchiectasis
* Pulmonary nodule requiring surgery
* History of recurrent respiratory infections (> 3 hospitalization in the last year)
* Clinically significant (> 4 Tablespoons per day) sputum production
* Fever, elevated white cell count, or other evidence of active infection
* Dysrhythmia that might pose a risk during exercise or training
* Congestive heart failure within 6 mo and LVEF < 45%
* Evidence or history of Cor Pulmonale
* Resting bradycardia (< 50 beats/min), frequent multifocal PVCs, complex ventricular arrhythmia, sustained SVT
* History of exercise-related syncope
* MI within 6 mo and LVEF < 45%
* Evidence of systemic disease or neoplasia expected to compromise survival during 5-yr period
* Any disease or condition that interferes with completion of initial or follow-up assessments
* Patient is currently enrolled in another clinical trial
* Patient is unable to complete 3 minutes of unloaded peddling on cycle ergometer
* Alpha-1-Antitrypsin Deficiency

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Mean % change in lung function (FEV1) | 90 days post index bronchoscopic lung volume reduction

SECONDARY OUTCOMES:
Mean % change in target lobe Residual Volume and Total Lung Capacity. Mean absolute change in dyspnea (mMRC-Score), Quality of life using St. George's Respiratory Questionnaire and SF-36. | 90 days post-index bronchoscopic lung volume reduction

CONTACTS AND LOCATIONS:
Overall Officials: Arschang Valipour, MD, Principal Investigator — Ludwig Boltzmann Institute for COPD
Locations (3):
- Otto Wagner Hospital, Vienna, Vienna, Austria
- Belgium (2):
  - University Antwerp, Antwerp
  - University Brussels, Brussels